CLINICAL TRIAL: NCT03405428
Title: Radial Artery Diameter Measurement By Ultrasonography For Determination Of Proper Cannula Size And Investigation Of Correlation Between Allen Test And Doppler Ultrasonography
Brief Title: Ultrasonography For Radial Artery Diameter Measurement And Its Correlation With Allen Test
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Guniz M.Koksal, Prof. Dr., Istanbul University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 419999
Record Dates: First submitted 2018-01-04; First posted 2018-01-23 (Actual); Last update posted 2018-03-13 (Actual); Status verified 2018-03

CONDITIONS: Anesthesia; Ultrasonography; Radial Artery; Catheterization
Keywords: Ultrasonography; Radial Artery Diameter; Allen Test; Arterial Cannulation; Doppler Ultrasonography; Ulnar Artery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- All patients (Other)
  Interventions: Other: Allen test; Other: Radial artery diameter measurement by ultrasonography; Other: Ulnar artery doppler ultrasonography

INTERVENTIONS:
Other: Allen test — Before induction, with firm occlusive pressure held on both the radial and ulnar arteries, the patient is asked to clench his or her fist several times until the palmar skin is blanched. The patient is then instructed to unclench the fist, and then ulnar artery pressure is released while maintaining occlusion of the radial artery. Overextension of the hand and wide spreading of the fingers should be avoided because it can lead to falsely abnormal results. The time required for palmar capillary refill is noted. An abnormal Allen test result was defined as a recovery time of more than 10 seconds.
Other: Radial artery diameter measurement by ultrasonography — Ultrasonography measurements will be performed with a linear probe before and after induction. The non-dominant hand of the patient will be fixed in the anatomical position on the arm chair. The wrist joint of patient will be extended to 30 degrees with a wrist pad. The USG probe will be transversally placed 2 cm proximal to the styloid process and the short axes of the radial artery will be scanned. The diameter of the radial artery will be measured and recorded.
Other: Ulnar artery doppler ultrasonography — Ultrasonography measurements will be performed with a linear probe before and after induction. The non-dominant hand of the patient will be fixed in the anatomical position on the arm chair. The wrist joint of patient will be extended to 30 degrees with a wrist pad. The USG probe will be transversally placed 2 cm proximal to the styloid process and the short axes of the ulnar arter will be scanned. The blood fow of ulnar artery will be measured and recorded.

SUMMARY:
In this study, the investigators will investigate how patients' radial artery diameters change according to sex, age, height, weight and body mass index by measuring radial artery diameter using ultrasonography. The correlation of Allen test with doppler ultrasonography will also be evaluated.

DETAILED DESCRIPTION:
Arterial catheterization for continuous hemodynamic monitoring or frequent blood sampling is a common procedure in anesthesia and critical care setting. The most commonly used site for arterial catheterization is the radial artery because of its superficial course, alternate blood supply to hand via ulnar artery and a low rate of complications. Allen test is a simple, but not reliable, method for assessing the safety of radial artery catheterization. Intraarterial catheterization has some complications such as hematoma, vasospasm, arterial thrombosis, necrosis of skin overlying. Using larger size cannula from radial artery diameter, increase rate of complications. The purpose of this study is to investigate the corelation of radial artery diameter with sex, age, height, weight and body mass index for determination of proper cannula size and investigation of correlation between Allen test and doppler ultrasonography.

ELIGIBILITY:
Inclusion Criteria:

* patients will be operated under general anesthesia
* patients were American Society of Anesthesiology (ASA) physical status I or II

Exclusion Criteria:

* ASA III, IV, V
* History of coroner artery disease
* History of peripheral artery disease,
* History of diabetes mellitus,
* History of hypertension
* Hemodynamic instability
* Hypovolemia
* History of Reynaud phenomenon
* History of hand or arm trauma
* previous catheterization

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 500 (Estimated)
Dates: Start 2018-02-01 (Actual); Primary Completion 2018-04-01 (Estimated); Study Completion 2018-04-30 (Estimated)

PRIMARY OUTCOMES:
change of the radial artery diameter according to sex, age, height, weight and body mass index | 5 minutes prior to anesthesia induction
  Ultrasonography measurements will be performed with a linear probe. The non-dominant hand of the patient will be fixed in the anatomical position on the arm chair. The wrist joint of patient will be extended to 30 degree with a wrist pad. The Ultrasonography probe will be transversally placed 2 cm proximal to the styloid process and the short axes of the radial artery will be scanned. The diameter of the radial artery will be measured and recorded.

SECONDARY OUTCOMES:
correlation between Allen test and doppler ultrasonography. | 5 minutes prior to anesthesia induction
  Before induction, with firm occlusive pressure held on both the radial and ulnar arteries, the patient is asked to clench his or her fist several seconds until the palmar skin is blanched. The patient is then instructed to unclench the fist, and then ulnar artery pressure is released while maintaining occlusion of the radial artery. The time required for palmar capillary refill is noted. An abnormal Allen test result was defined as a recovery time of more than 10 seconds. Ultrasonography measurements will be performed with a linear probe. The non-dominant hand of the patient will be fixed in the anatomical position on the arm chair. The wrist joint of patient will be extended to 30 degree with a wrist pad. The USG probe will be transversally placed 2 cm proximal to the styloid process and the short axes of the ulnar artery will be scanned. The blood fow of ulnar artery will be measured and recorded.
change of the radial artery diameter according to sex, age, height, weight and body mass index after the induction | 5 minutes following to anesthesia induction
  Ultrasonography measurements will be performed with a linear probe. The non-dominant hand of the patient will be fixed in the anatomical position on the arm chair. The wrist joint of patient will be extended to 30 degree with a wrist pad. The USG probe will be transversally placed 2 cm proximal to the styloid process and the short axes of the radial arter will be scanned. The diameter of the radial artery will be measured and recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Güniz Meyancı Köksal, Prof., Principal Investigator — Istanbul University Cerrahpasa Medical Faculty
Locations (1):
- Istanbul University Cerrahpasa Medical Faculty, Istanbul, Turkey (Türkiye)